CLINICAL TRIAL: NCT05384275
Title: Aerosol Generation After Tracheal Extubation With High-flow Nasal Oxygen Therapy Compared With Standard Low-flow Oxygen Therapy: a Randomised Controlled Trial
Brief Title: High-Flow Aerosol Generation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P02723
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Oxygen Therapy; Heart Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention: Standard Oxygen Therapy (No Intervention): Standard oxygen therapy arm patients will be given 30-40% inspired O2 and flow 2-6 l/min via nasal prongs or non-rebreathing mask (not humidified and not heated) post extubation. Monitoring of saturations, respiratory rate and arterial gases will happen 15 minutes post extubation and then as per local policy thereafter. If saturations < 93% then FiO2 will be increased as per respiratory escalation protocol. Standard oxygen therapy will be given for a minimum of 16 hours post extubation.
- High-Flow Nasal Therapy (Active Comparator): High-flow nasal therapy arm patients will be given AIVRO 2 high flow oxygen therapy machines post extubation, start at 30-40% inspired O2 and flow 30 l/min then up to 50 l/min over 5-10 min. Monitoring of saturations, respiratory rate and arterial gases will happen after 15 minutes post extubation and then as per local policy thereafter. If saturations < 93% then increase FiO2 as per respiratory escalation protocol. High flow nasal therapy will be given for a minimum of 16 hours post extubation.
  Interventions: Device: High Flow Nasal Therapy

INTERVENTIONS:
Device: High Flow Nasal Therapy — High Flow Nasal Oxygen (Airvo2 Device)
  Arms: High-Flow Nasal Therapy

SUMMARY:
The study will be measuring aerosol generated from the point of tracheal extubation after cardiac surgery in patients who then receive either high-flow nasal oxygen therapy (HFNT) or standard low-flow oxygen therapy, who have been consented to participate within another randomised controlled trial (The NOTACS Study, IRAS ID 278290). Aerosol generation will be compared at various sizes of particles < 10 microns in size and sampled in different locations in the standardised patient care rooms in the ICU. The rate of change of aerosol generation, maximum aerosol generation and duration of aerosol production greater than background will be investigated. The aim is to compare high-flow and standard low-flow oxygen therapy to determine if there is a difference in aerosol generation between the therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over.
2. Undergoing elective or urgent first-time or redo cardiac surgery (CABG, valve surgery, surgery on the aorta or any combination).
3. Have one or more clinical patient-related risk factor for postoperative pulmonary complications (COPD, asthma, lower respiratory tract infection in last 4 weeks as defined by use of antibiotics, body mass index ≥35 kg/m2, current (within the last 6 weeks) heavy smokers (> 10 pack years))(26, 27).

For the purposes of the study, the following definitions apply:

Asthma is a disease characterized by recurrent attacks of breathlessness and wheezing, and patients will have been prescribed medication by inhalers or nebulisers (either bronchodilators or steroids).

Chronic Obstructive Pulmonary Disease (COPD) is an umbrella term used to describe chronic lung diseases that cause limitations in lung airflow. The more familiar terms 'chronic bronchitis' and 'emphysema' are no longer used but are now included within the COPD diagnosis. The most common symptoms of COPD are breathlessness, or a 'need for air', excessive sputum production, and a chronic cough. Patients suitable for the NOTACS study will have been prescribed medication by inhalers or nebulisers (either bronchodilators or steroids).

Exclusion Criteria:

1. Requiring home oxygen therapy.
2. Deep hypothermic circulatory arrest planned.
3. Contraindication to HFNT, e.g. nasal septal defect.
4. Requirement for home respiratory support (including: CPAP, BiPAP).
5. Requiring emergency cardiac surgery defined as surgery required within 24 hours of the decision to operate.
6. Patient's not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
To assess aerosol generation as measured by total exposure level of 0.3 micron particles during tracheal extubation and for 1 hour afterwards (study period) at 50 cm to the side of the patient's head. | 1 hour
  This will be measured by the total particle count using area under the curve (AUC) over the 1 hour timeframe.

SECONDARY OUTCOMES:
To assess the time needed for particle counts to return to baseline level, measuring particles size 0.3, 0.5, 1.0, 2.5, 5.0 and 10.0 microns during tracheal extubation and for 1 hour afterwards. | 1 hour
  Measured at 50 cm to the side of the patient's head, at 50 cm from the top of the patient's head and by the patient's feet.
To assess total aerosol generation measuring particles size 0.5, 1.0, 2.5, 5.0 and 10.0 microns during tracheal extubation and for 1 hour afterwards. | 1 hour
  Measured at 50 cm to the side of the patient's head, at 50 cm from the top of the patient's head and by the patient's feet.
To assess total aerosol generation measuring particle size 0.3 microns during tracheal extubation and for 1 hour afterwards at 50 cm from the top of the patient's head and by the patient's feet. | 1 hour
To assess the peak particle count of 0.3, 0.5, 1.0, 2.5, 5.0 and 10.0 micron during tracheal extubation and for 1 hour afterwards at 50 cm to the side of the patient's head, 50 cm from the top of the patient's head and by the patient's feet. | 1 hour
To measure CO2 levels during tracheal extubation and for 1 hour afterwards. | 1 hour
  Measured at 50 cm to the side of the patient's head, at 50 cm from the top of the patient's head and by the patient's feet. A CO2 counter will be placed next to each of the particle counter devices.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Klein, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No